CLINICAL TRIAL: NCT00365001
Title: A Randomized, Open-label Study to Assess the Pharmacokinetics of Simvastatin and Methotrexate in Combination With Tocilizumab in Patients With Rheumatoid Arthritis.
Brief Title: A Drug Interaction Study Between Tocilizumab, Methotrexate and Simvastatin on Patients With Rheumatoid Arthritis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Clinical Trials, Study Director, Hoffmann-La Roche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WP18663
Record Dates: First submitted 2006-08-15; First posted 2006-08-16 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Methotrexate; Simvastatin

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]; Drug: Methotrexate; Drug: Simvastatin
- 2 (Active Comparator)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]; Drug: Methotrexate

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 10mg/kg iv on day 8
Drug: Methotrexate — 10-25mg po/week
Drug: Simvastatin — 40mg po on days 1, 15 and 43
  Arms: 1

SUMMARY:
This 2 arm study will investigate the pharmacokinetics of simvastatin and methotrexate in combination with tocilizumab to assess any potential drug interactions. Patients will be randomized to receive either tocilizumab (10mg/kg iv infusion on day 8) + methotrexate (10-25mg po /week) or tocilizumab + methotrexate + simvastatin (40mg po on days 1, 15 and 43). Blood samples will be taken for analysis at intervals up to day 44. The anticipated time on study treatment is <3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* rheumatoid arthritis for >=6 months;
* methotrexate for >=12 weeks prior to day 1 (stable at 10-25mg/week for 8 weeks).

Exclusion Criteria:

* history of, or current inflammatory joint disease or rheumatic autoimmune disease other than RA;
* concurrent treatment with any DMARD other than methotrexate;
* prior treatment with tocilizumab.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters for simvastatin and metabolite, and methotrexate and metabolite. | Days 1, 15 and 43

SECONDARY OUTCOMES:
Pharmacokinetic parameters for tocilizumab. | Days 11, 22, 29 and 36.
CRP, IL-6, sIL-6R changes | Throughout study
AEs, laboratory parameters. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- United States (10):
  - Anniston, Alabama
  - Scottsdale, Arizona
  - Little Rock, Arkansas
  - Jacksonville, Florida
  - Palm Harbor, Florida
  - Royal Oak, Michigan
  - Omaha, Nebraska
  - Oklahoma City, Oklahoma
  - Duncansville, Pennsylvania
  - Austin, Texas
- Christchurch, New Zealand

REFERENCES:
- [Derived] Schmitt C, Kuhn B, Zhang X, Kivitz A, Grange S. Tocilizumab has no clinically relevant effects on methotrexate pharmacokinetics in patients with rheumatoid arthritis. Int J Clin Pharmacol Ther. 2012 Mar;50(3):218-23. doi: 10.5414/cp201613. PMID 22373834